CLINICAL TRIAL: NCT03167307
Title: OMEGA-3 FATTY ACIDS AS FIRST-LINE TREATMENT IN PAEDIATRIC DEPRESSION. A Phase III, 36-week, Multi-centre, Double-blind, Placebo-controlled Randomized Superiority Study
Brief Title: The Omega-3 Fatty Acid Paediatric Depression Trial
Acronym: Omega-3-pMDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gregor Berger (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Gregor Berger, Head of Developmental Psychopharmacology Group, Department of Child and Adolescent Psychiatry, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNF 33IC30_166826; 2016-02116 (Other: Swissethics)
Record Dates: First submitted 2017-02-24; First posted 2017-05-25 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Depression
Keywords: omega-3 fatty acids; eicosapentaenoic acid; docosahexaenoic acid; antidepressants; suicidality; cognition; childhood depression; pediatric depression
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — Fatty Acids, Omega-3; Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: A 36-week, multi-centre, double-blind, placebo-controlled randomized superiority Study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 fatty acid oil (Experimental): A daily dose of 500mg EPA/ 250mg DHA in the 8 to <13 year olds, and 1000mg EPA / 500mg DHA in the 13 to <18 years olds, respectively, will be added to standardized treatment according to the German S3 Guidelines for the treatment of depression in children and adolescents
  Interventions: Drug: Omega 3 fatty acid
- Placebo oil (Placebo Comparator): Placebo capsules will contain mostly medium chain triglycerides (MCT) and also a small amount of fish oil to mimic the fishy flavour and taste. Placebo will be added to standardized treatment according to the German S3 Guidelines for the treatment of depression in children and adolescents
  Interventions: Drug: Placebo oil

INTERVENTIONS:
Drug: Omega 3 fatty acid — Omega-3 fatty acids in addition to standard treatment for depression in children and adolescents according to the German S3 Guidelines
  Other Names: Eicosapentaenoic acid (EPA) / docosahexaenoic acid (DHA)
  Arms: Omega-3 fatty acid oil
Drug: Placebo oil — medium chain triglycerides in addition to standard treatment for depression in children and adolescents according to the German S3 Guidelines
  Other Names: medium chain triglycerides
  Arms: Placebo oil

SUMMARY:
This study investigates the therapeutic efficacy and safety of omega-3 fatty acids rich in eicosapentaenoic acid / docosahexaenoic acid in pediatric depression in a nine months double-blind multi-centre study in 220 children and adolescents between 8 and 17 years of age. Inflammatory and bioactive lipid markers as predictors of response are evaluated. The relationship between omega-3 fatty acids with psychopathology, illness course and cognitive parameters will be further investigated.

DETAILED DESCRIPTION:
Background: About 10% teenagers report moderate to marked depressive symptoms and between 1-6% will develop a paediatric major depressive disorder (pMDD) until adulthood. However, evidence-based treatment approaches are sparse and the use of selective serotonin reuptake inhibitors (SSRIs) is heavily debated due to reports of an increase in suicidal ideation and limited efficacy in this age group. Growing evidence suggests that omega-3 fatty acids may be a beneficial treatment in adult MDD (aMDD) with no published study in teenagers, despite of its face validity as a valuable first-line treatment. Meta-analyses of published randomized controlled trials (RCTs) in aMDD show moderate effect sizes, if the proportion of eicosapentaenoic acid (EPA) is >60% of the total omega-3 fatty acids. One small RCT in prepubertal children shows an even larger effect size in favour of omega-3 fatty acids. Higher inflammatory mediators (e.g. c-reactive protein, interleukins and others) have been reported in aMDD and pMDD. Preliminary data suggests that a proinflammatory state may serve as predictor for omega-3 fatty acids response. Furthermore, low levels of omega-3 fatty acids have been found in aMDD and pMDD potentially also serving as EPA-response predictors. As MDD is a heterogeneous disease entity, such response predictors should be incorporated into MDD RCTs.

Objective: 1) To investigate the therapeutic efficacy and safety of omega-3 fatty acids rich in EPA in pMDD, 2) to demonstrate clinical meaningful effects of omega-3 fatty acid treatment, 3) to investigate inflammatory and bioactive lipid markers as response predictors, and 4) to investigate the relationship between psychopathology (in particular suicidal ideation), illness course and cognition in relation to inflammatory and bioactive lipid markers. 5.) To establish a tissue repository of phenotypically well characterised children and adolescents with pMDD.

Outcome: The German S3 Guidelines for the treatment of depression in children and youth define the background treatment for all participants. All clinical partners will be trained and monitored accordingly. The primary outcomes are the (continuous) Children's Depression Rating Scale-revised (CDRS-R) total score and the (dichotomous) rates of recovery defined by the absence of pMDD for >4months at 36 weeks, as well as response and remission rates at 12 and 36 weeks. Inflammatory mediators in serum using immunoassays, red blood cell omega-3, 6, 9 and trans fatty acids using gas chromatography (GC) and bioactive lipid mediators (e.g. E-series resolvin) using mass spectrometry (LC-MS/MS) will be measured as potential response predictors. Adverse events/ harm endpoints (in particular suicidality) will be coded using MedDRA. Adherence measurements are pill counts, as well as n-3 EPA/DHA levels across the study. Blood samples will be taken at study entry, week 12 and 36.

Study design:A Swiss, multicentre, randomised, double-blind, placebo-controlled clinical trial.

Inclusion / Exclusion criteria:The study aims to recruit a sample of 220 individuals aged 8 -17 years, who are in- or outpatients of a participating centre and have a present primary diagnosis of major depressive disorders with depressive symptom of at least moderate severity. Participants with pre-existing neurological or medical conditions likely to be responsible for the depressive symptoms or other psychopathological diagnoses are excluded.

Measurement and procedures: The study design incorporates a 1-2week screening, a 1-week lead-in and a 36-week double-blind placebo-controlled treatment phase. The severity of the depression and psychosocial functioning will be assessed at baseline and at each study visit (twice in the acute phase and twice in the maintenance phase) using a variety of different questionnaires and rating scales. Cognitive testing and biological markers (blood, urine and saliva) will be sampled at baseline and at 12 and 36 weeks. Adherence to the study will be checked by pill count at each study visit and polyunsaturated fatty acid (PUFA) level measurements in red blood cell membranes at baseline, 12 and 36 weeks will be performed.

Study product / Intervention: In the proposed study a daily dose of 500mg EPA/ 250mg DHA in the 8 to <13 year olds and 1000mg EPA / 500mg DHA in the 13 to <18 years olds (which corresponds with the omega-3 fatty acid doses used in adult MDD RCTs) is used as an active treatment, respectively. The drug will be administered for 36 weeks. Placebo capsules will contain mostly medium chain triglycerides (MCT) and also a small amount of fish oil to mimic the fishy flavour and taste. All study medication (active and placebo) will use fish derived gelatine capsules and natural orange flavor.

Sample size justification: This clinical trial aims to include 220 participants in total, resulting in 110 participants per treatment group. A sample size calculation was performed based on the effect size of 0.54 found in a previous meta-analysis on the effect of omega-3 fatty acids in aMDD. Sample size calculations were then adjusted for an expected higher placebo-response rate in minors and given the multi-centre design. The analysis resulted that the inclusion of 108 patients per treatment group will achieve 80% or greater power to detect a difference of 20% in response rates between the two treatment groups. The sample of 220 participants exceeds therefore the projected sample size needed to detect a clinical meaningful difference. Participants with no psychopathological follow up data at all will be replaced.

Study duration: The study duration is projected to be about four years and (April 2017 - 2021) for patient recruitment and assessment and another year to finish up all the analysis and generate the final study report.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in- or outpatients of a participating centre
* Children aged 8 <13 years or teenager aged 13 to < 18 years
* Major depressive disorder with depressive symptoms of at least moderate severity
* Written informed consent of the parents / legal representatives and patients' assent

Exclusion Criteria:

* contraindications to the drug
* more than 4 weeks of regular omega-3 supplementation
* pregnant or breastfeeding or intention to become pregnant
* pre-existing neurological or medical conditions likely to be responsible for depressive symptoms
* laboratory screening values considered clinically relevant
* known or suspected non-compliance
* other psychiatric diagnoses (substance dependency, schizophrenia, bipolar affective disorder, eating disorder, mental retardation, pervasive developmental disorder)
* inability to follow the procedures of the study
* Participation in another study with omega-3, previous enrolment in the current study, or dependent persons of the investigators

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 257 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Symptomatic improvement | 9 months
  Change of the (continuous) Children's Depression Rating Scale-revised (CDRS-R) total score analyzed using using a linear random coefficient regression model

SECONDARY OUTCOMES:
Response rate | 6 weeks
  Response is defined as a 30% decrease in total baseline CDRS sum score
Remission rate | 9 months
  remission is defined as a CDRS total score <28
Scale of Impulsivity and Emotion Dysregulation (IES-27) | 9 months
  Correlation between omega-3 index and the overall score of the Scale of Impulsivity and Emotion Dysregulation (IES-27)
Antidepressant medication | 9 months
  Differences in antidepressant medication between the treatment groups
Children's global assessment scale (CGAS) | 9 months
  Differences in the scores of the CGAS between treatment groups
Kidscreen quality of life measure for children and adolescents | 9 months
  Differences in the scores of the Kidscreen between treatment groups
Hospitalization | 9 months
  Differences in hospital admissions between the treatment groups
Retention rate | 9 months
  Differences in retention rate between the treatment groups
Inflammatory mediators as predictors of response | Baseline values as predictors for response across the trial
  Omega-3 fatty acid response wil be predicted by the ratio between pro- and anti-inflammatory markers
Metabolites of EPA as predictors for response | Baseline values as predictors for response across the trial
  Omega-3 fatty acid response will be predicted by the levels of direct metabolites of EPA
Omega-3 index as predictors of response | Baseline values as predictors for response across the trial
  Omega-3 fatty acid response will be predicted by the omega-3 index
Depressive Symptoms | 9 months
  Correlation between severity of depressive symptoms and pro-inflammatory state and omega-3 index
Suicidal ideation Questionnaire (SIQ) | 9 months
  Inverse correlation between omega-3 fatty acids and scores in the SIQ
Relationship between stress, omega-3 fatty acids and saliva cortisol | 9 months
  Correlation between omega-3 fatty acid levels, scores in the perceived stress scale and saliva cortisol
Recovery rate | 9 months
  (dichotomous) rates of recovery defined by the absence of pMDD for >4months at 36 weeks according to the Kiddie-Schedule (K-SADS)
Remission rate | 3 months
  remission is defined as a CDRS total score <28

OTHER OUTCOMES:
Verbal learning and memory test (VLMT) | 9 months
  Differences in the overall score between the treatment groups
Behavior Rating Inventory of Executive Function (BRIEF) | 9 months
  Differences in the scores of the BRIEF between the treatment groups
Tolerability assessed by the Self-reported Antidepressant Side-Effect Checklist (ASEC) | 9 months
  ASEC total score shows no significant differences between active and placebo
Digit span measured by the Wechsler Intelligence Scale for Children (WISC-IV) | 9 months
  Differences in the overall score of the digit span between the treatment groups
Emotion recognition measured with the Amsterdam Neuropsychological Task (ANT) Program | 9 months
  Significant better scores in emotion recognition of the active compared to the placebo group
Attentional flexibility measured with the shifting attentional set of the Amsterdam Neuropsychological Task (ANT) program | 9 months
  Differences in the reaction times between the treatment groups
Regensburg Word Fluency Test (RWT) | 9 months
  Differences in the number of generated words in the RWT between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Walitza, MD, Principal Investigator — Psychiatrische Universitätsklinik Zürich KJPP; Klaus Schmeck, MD, Principal Investigator — Universitäre Psychiatrische Kliniken (UPK) Basel
Locations (7):
- Switzerland (7):
  - Psychiatric Services Baselland, Liestal, Basel-Landschaft
  - Psychiatric University Clinics, Department of Child and Adolescent Psychiatry, Zurich, Canton of Zurich
  - Klinik Sonnenhof, Ganterschwil, St.Gallen
  - Clienia Littenheid, Littenheid, Thurgau
  - Spital Thurgau Kinder- und Jugendpsychiatrischer Dienst, Weinfelden, Thurgau
  - University Psychiatric Services, Basel
  - Stiftung Kinder- und Jugendpsychiatrische Dienste St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
A BioBank will be established. Access to the Biobank can be requested upon completion of the trial contacting the sponsor-investigator Dr. Gregor Berger

REFERENCES:
- [Derived] Berger G, Haberling I, Emery S, Albermann M, Baumgartner N, Nalani K, Strumberger M, Wockel L, Erb S, Bachmann S, Muller-Knapp U, Contin-Waldvogel B, Yamini A, Rhiner B, Drechsler R, Held U, Reeve K, Heinz P, Pauli D, Schmeck K, Hersberger M, Walitza S; Omega-3 pMDD Study Group. omega-3 Fatty Acids in Pediatric Major Depressive Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2548703. doi: 10.1001/jamanetworkopen.2025.48703. PMID 41481294
- [Derived] Preisig M, Haberling I, Smigielski L, Emery S, Baumgartner N, Albermann M, Strumberger M, Schmeck K, Wockel L, Erb S, Rhiner B, Contin-Waldvogel B, Walitza S, Berger G. The mediating role of depression in the association between health-related quality of life and suicidal ideation in adolescents: findings from a longitudinal study. Front Child Adolesc Psychiatry. 2025 Aug 14;4:1567387. doi: 10.3389/frcha.2025.1567387. eCollection 2025. PMID 40894517
- [Derived] Haberling I, Preisig M, Emery S, Baumgartner N, Albermann M, Strumberger M, Schmeck K, Wockel L, Erb S, Rhiner B, Contin B, Walitza S, Berger G. Clinical characteristics of depressed children and adolescents with and without suicidal thoughts and behavior: a cross-sectional study. Front Child Adolesc Psychiatry. 2025 Feb 21;4:1510961. doi: 10.3389/frcha.2025.1510961. eCollection 2025. PMID 40061518
- [Derived] Albermann M, Emery S, Baumgartner N, Strumberger M, Erb S, Wockel L, Muller-Knapp U, Rhiner B, Contin-Waldvogel B, Bachmann S, Schmeck K, Berger G; Omega-3 Study Team; Haberling I. Executive functions and borderline personality features in adolescents with major depressive disorder. Front Hum Neurosci. 2023 Jun 22;17:957753. doi: 10.3389/fnhum.2023.957753. eCollection 2023. PMID 37425294
- [Derived] Haberling I, Berger G, Schmeck K, Held U, Walitza S. Omega-3 Fatty Acids as a Treatment for Pediatric Depression. A Phase III, 36 Weeks, Multi-Center, Double-Blind, Placebo-Controlled Randomized Superiority Study. Front Psychiatry. 2019 Nov 27;10:863. doi: 10.3389/fpsyt.2019.00863. eCollection 2019. PMID 31827448
- See also: Study website (online from Mai 2017) — https://www.omega3.uzh.ch

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Original version (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03167307/Prot_SAP_000.pdf
  • Study Protocol: Final version (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03167307/Prot_001.pdf
  • Statistical Analysis Plan: detailled statistical analysis plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03167307/SAP_002.pdf